CLINICAL TRIAL: NCT02662218
Title: Prospective, Multicenter, Observational Study to Evaluate the Clinical Performance of a Sterile, Bacteria-binding, Super-absorbent Wound Dressing
Brief Title: Observational Study of Clinical Performance of a Sterile, Bacteria-binding, Super-absorbent Wound Dressing
Status: Completed | Type: Observational
Sponsor: BSN Medical GmbH (Industry)
Responsible Party: Sponsor
Other Study IDs: C1438
Record Dates: First submitted 2016-01-08; First posted 2016-01-25 (Estimated); Last update posted 2017-06-21 (Actual); Status verified 2017-06

CONDITIONS: Wounds
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with superficial wounds: A cohort of 50 patients with superficial wounds of any etiology (see inclusion criteria), who need advanced wound care treatment in any case, will be observed over a period of 14 days; the exact duration for each patient depends upon the investigator's assessment. The observation consists of an initial visit, at least one dressing change after max. 7 days and a final visit. Patients will be treated with the CE-marked wound care product. This product is already in general use in the Netherlands and Germany. It is a sterile, bacteria-binding, super-absorbent wound dressing. Apart from the predefined study visits, daily dressing changes in accordance with daily clinical practice are possible.

SUMMARY:
This prospective, multicenter, single-arm observational study aims to document the clinical performance and safety of a sterile, bacteria-binding, super-absorbent wound dressing for the intended use in a daily clinical practice. 50 patients (male/female) with superficial wounds of any etiology affecting only epidermis and dermis layer, with one or more clinical signs of infection or at high risk of infection and also high to very high exudate levels will be observed over a period of 14 days.

ELIGIBILITY:
Inclusion Criteria:

* Men and women ≥ 18 years old
* Written informed consent after patient education to participate in the study
* Superficial wounds of any etiology affecting only epidermis and dermis layers
* Maximum wound size: 6 x 16cm / 6 x 6cm
* Wounds with one or more clinical signs or infection or assessed as at high risk of infection according to the following:

  * Wounds assessed as critically colonized with malodour, abnormal tissue or absence of viable tissue, excessive or increased serous exudate, possible extension of wound dimensions and no sign of a healing process and/or
  * Wounds with one or more historical episodes of topical infection and/or
  * Wounds assessed as at a high risk of infection on other grounds by the investigator.
* Superficial wounds with high levels of exudate

Exclusion Criteria:

* Not willing to sign or incapable of signing an informed consent form
* Known allergy or sensitivity to one of the dressing components
* Pregnancy or lactation
* Subject is participating in another clinical study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with superficial wounds of any etiology, that are treated at outpatients' clinic
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Number of patients with persisting infections will be documented in a standardized Case Report Form (CRF). | 14 days
  Symptoms such as odor, pain, localized heat and erythema will be assessed by a clinician and documented in four different categories depending on its severity.
Number of participants with newly developed infections will be documented in a standardized Case Report Form (CRF) | 14 days
  Symptoms such as odor, pain, localized heat and erythema will be assessed by a clinician and documented in four different categories depending on its severity.

CONTACTS AND LOCATIONS:
Overall Officials: Nicky Ivins, Principal Investigator — Welsh Wound Innovation Centre
Locations (1):
- Welsh Wound Innovation Centre, Ynysmaerdy, Rhondda Cynon Taf, United Kingdom